CLINICAL TRIAL: NCT06071377
Title: Achieving Understanding of the Natural History of Sickle Cell Trait (AUNT)
Status: Recruiting | Type: Observational
Sponsor: National Alliance for Sickle Cell Centers (Other)
Collaborators: Beam Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AUNT
Record Dates: First submitted 2023-09-26; First posted 2023-10-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Trait
MeSH Terms: conditions — Sickle Cell Trait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For individuals who consent to provide optional DNA testing, an alpha globin sequencing (ATHAL) test will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with sickle cell trait
  Interventions: Other: Biologic Specimen Collection

INTERVENTIONS:
Other: Biologic Specimen Collection — Participants will have blood and urine collected at Baseline

SUMMARY:
The main purpose of this study is to create a longitudinal cohort of those with Sickle Cell Trait (SCT) to better understand the hematologic phenotype for those that carry HbS, assess for differences in those with varying quantities of HbS and assess for potential clinical complications of SCT.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing to voluntarily participate and sign the study consent
2. Know/suspect they have SCT and are willing to get tested to confirm/learn about their SCT status
3. Adults ages 18 and older

Exclusion Criteria:

1. Unwilling to sign consent
2. Known end-stage renal disease or dialysis
3. Known SCD (including sickle cell-beta thalassemia)
4. People who do not have SCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 and older with sickle cell trait.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin variant quantification | Through study completion, an average of 2 years
  Determine range of variability in baseline %HbS in SCT subjects and relationship of baseline %HbS to markers of hemolysis (LDH, reticulocytes, haptoglobin), coagulopathy (D-dimer), and renal disease (urine albumin/creatinine ratio)

SECONDARY OUTCOMES:
Red blood cell rheology | Through study completion, an average of 2 years
  Identify range of variation in baseline RBC rheological parameters in SCT subjects and relationship to %HbS, other baseline clinical parameters
Natural History | Through study completion, an average of 2 years
  Evaluate the frequency of hemolysis
  * Evaluate potential for and progression of chronic kidney disease and albuminuria
  * Evaluate the relative risk of thrombosis based on medical history
  * Evaluate the prevalence of episodes of pain or exercise-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Julie Kanter, MD, Principal Investigator — National Alliance for Sickle Cell Centers
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - Loma Linda University Health Care, Loma Linda, California
  - Nemours Children's Hospital, Wilmington, Delaware
  - Indiana University, Indianapolis, Indiana
  - Functional Fluidics, Detroit, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - UT Health Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No